CLINICAL TRIAL: NCT04905979
Title: Randomized Double-Blind 2-Period Multiple Dose Crossover Study to Evaluate the Efficacy and Safety of AD113 vs Atomoxetine in OSA Patients With Hypertension
Brief Title: Trial of AD113 and Atomoxetine in OSA Patients With Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apnimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APX-002
Record Dates: First submitted 2021-05-20; First posted 2021-05-28 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-03

CONDITIONS: Obstructive Sleep Apnea; Hypertension
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AD113 (Experimental): Two oral capsules administered before bed
  Interventions: Drug: AD113
- Atomoxetine (Experimental): Two oral capsules administered before bed
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: AD113 — Two oral capsules administered before bed
  Arms: AD113
Drug: Atomoxetine — Two oral capsules administered before bed
  Arms: Atomoxetine

SUMMARY:
This is a randomized, double blind, 2-period, non placebo-controlled crossover study in patients with moderate to severe OSA and controlled hypertension, comparing atomoxetine with AD113

DETAILED DESCRIPTION:
The study is designed to examine the efficacy and safety of AD113 to treat obstructive sleep apnea with hypertension. The study is a two-period multi-dose randomized crossover design in which patients will undergo overnight polysomnographic (PSG) testing with dosing of one of the following 2 treatments: AD113 for 10 days or Atomoxetine for 10 days. Participants will return 1 week after their final crossover PSG for an end of study (EOS) Visit.

ELIGIBILITY:
Inclusion Criteria:

* Between 25 to 65 years of age, inclusive, at the Screening Visit.
* AHI 10 to 50 (hypopneas defined by 4% oxygen desaturation)
* History of hypertension or blood pressure at Visit 1 ≥130/80 mmHg

Exclusion Criteria:

* History of narcolepsy.
* Clinically significant craniofacial malformation.
* Clinically significant cardiac disease (e.g., rhythm disturbances, coronary artery disease or cardiac failure) or hypertension requiring more than 2 medications for control. A medication for these purposes is defined by dosage form, such that a combination antihypertensive medication is considered 1 medication
* CPAP should not be used for at least 2 weeks prior to first study PSG
* History of using oral or nasal devices for the treatment of OSA may enroll as long as the devices are not used during participation in the study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-07-31 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change in hypoxic burden (HB, total area under the respiratory event-related desaturation curve) | 10 days of treatment per crossover arm
  Change in HB for AD113 vs. atomoxetine measured by polysomnography atomoxetine

SECONDARY OUTCOMES:
Change in Apnea-Hypopnea Index (AHI, average number of events for every hour of sleep) | 10 days of treatment per crossover arm
  Change in AHI for AD113 vs. atomoxetine measured by polysomnography

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - PCCAB, Towson, Maryland
  - Intrepid Research, Cincinnati, Ohio
  - Bogan Sleep Consultants, Columbia, South Carolina

REFERENCES:
- [Derived] Schwartz AR, Herpel L, Bogan R, Corser B, Pho H, Taranto-Montemurro L. Atomoxetine and spironolactone combine to reduce obstructive sleep apnea severity and blood pressure in hypertensive patients. Sleep Breath. 2024 Dec;28(6):2571-2580. doi: 10.1007/s11325-024-03113-1. Epub 2024 Sep 21. PMID 39305436